CLINICAL TRIAL: NCT06391840
Title: Airway Ultrasound As an Independent Predictor of Difficult Laryngoscopy in Patients Receiving General Anesthesia for Elective Surgery
Status: Recruiting | Type: Observational
Sponsor: DIMITRIOS KATSAROS (Other)
Responsible Party: Sponsor-Investigator, DIMITRIOS KATSAROS, Dimitrios Katsaros, MD, G.Gennimatas General Hospital
Organization: G.Gennimatas General Hospital (Other)
Other Study IDs: GGennimatasGH 18418
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-04

CONDITIONS: Airway Ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients listed for elective surgery
  Interventions: Other: Airway ultrasound

INTERVENTIONS:
Other: Airway ultrasound — Pre-operative airway ultrasound

SUMMARY:
The goal of this observational study is to determine the usefulness of pre-operative airway ultrasound in predicting difficult laryngoscopy in patients receiving general anesthesia for elective surgery. The main question it aims to answer is the independent prognostic value of pre-operative airway ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* listed for elective surgery
* airway assessment is possible prior to anesthesia

Exclusion Criteria:

* refusal to be enrolled in study
* airway assessment is not possible prior to anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients above 28 years of age listed for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Independent prognostic value of airway ultrasound in difficult laryngoscopy | Airway assessment prior to anesthesia, usually 1-2 days before. Statistical analysis will be conducted after all data has been gathered

SECONDARY OUTCOMES:
Search of normal and pathological values in airway ultrasound measurements | Airway assessment prior to anesthesia, usually 1-2 days before. Statistical analysis will be conducted after all data has been gathered

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Katsaros, Principal Investigator — G.Gennimatas General Hospital
Locations (1):
- G. Gennimatas General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carsetti A, Sorbello M, Adrario E, Donati A, Falcetta S. Airway Ultrasound as Predictor of Difficult Direct Laryngoscopy: A Systematic Review and Meta-analysis. Anesth Analg. 2022 Apr 1;134(4):740-750. doi: 10.1213/ANE.0000000000005839. PMID 34914641
- [Background] You-Ten KE, Siddiqui N, Teoh WH, Kristensen MS. Point-of-care ultrasound (POCUS) of the upper airway. Can J Anaesth. 2018 Apr;65(4):473-484. doi: 10.1007/s12630-018-1064-8. Epub 2018 Jan 18. PMID 29349733
- [Background] Adi O, Fong CP, Sum KM, Ahmad AH. Usage of airway ultrasound as an assessment and prediction tool of a difficult airway management. Am J Emerg Med. 2021 Apr;42:263.e1-263.e4. doi: 10.1016/j.ajem.2020.09.011. Epub 2020 Sep 14. PMID 32994082
- [Background] Osman A, Sum KM. Role of upper airway ultrasound in airway management. J Intensive Care. 2016 Aug 15;4:52. doi: 10.1186/s40560-016-0174-z. eCollection 2016. PMID 27529028
- [Background] Xu J, Wang B, Wang M, Yao W, Chen Y. The value of multiparameter combinations for predicting difficult airways by ultrasound. BMC Anesthesiol. 2022 Oct 5;22(1):311. doi: 10.1186/s12871-022-01840-0. PMID 36199026
- [Background] Gottlieb M, Holladay D, Burns KM, Nakitende D, Bailitz J. Ultrasound for airway management: An evidence-based review for the emergency clinician. Am J Emerg Med. 2020 May;38(5):1007-1013. doi: 10.1016/j.ajem.2019.12.019. Epub 2019 Dec 11. PMID 31843325